CLINICAL TRIAL: NCT01181141
Title: A Phase 3, Randomized, Open Label, Safety and Efficacy Study of the Oral Factor Xa Inhibitor DU-176b Compared With Enoxaparin Sodium for Prevention of Venous Thromboembolism in Patients After Hip Fracture Surgery (STARS J-4 Trial)
Brief Title: Study of DU-176b, Prevention of Venous Thromboembolism in Patients After Hip Fracture Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DU176b-B-J303
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2015-02

CONDITIONS: Venous Thromboembolism
Keywords: Anticoagulants; Enoxaparin sodium; venous thromboembolism.; thromboembolism; Thrombosis; deep vein thrombosis; DU-176b; Edoxaban; factor Xa; hip fracture surgery; embolism
MeSH Terms: conditions — Venous Thromboembolism; Thromboembolism; Thrombosis; Venous Thrombosis; Embolism | interventions — edoxaban; enoxaparin sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DU-176b (Experimental): DU-176b oral tablets, 30 mg., taken once daily for 2 weeks, initiated within 6 to 24 hours after surgery
  Interventions: Drug: DU-176b (edoxaban)
- Enoxaparin sodium (Active Comparator): Enoxaparin sodium 20mg(=2000IU)/0.2ml twice daily, subcutaneous injection for 2 weeks, initiated within 24 to 36 hours after surgery
  Interventions: Drug: Enoxaparin sodium 20mg

INTERVENTIONS:
Drug: DU-176b (edoxaban)
  Arms: DU-176b
Drug: Enoxaparin sodium 20mg
  Arms: Enoxaparin sodium

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of DU-176b compared with enoxaparin sodium for the prevention of venous thromboembolism in patients after elective hip fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are scheduled to undergo surgery within 10 days for fracture of inner or outer femoral neck (trochanteric and subtrochanteric)

Exclusion Criteria:

* Subjects with risks of hemorrhage
* Subjects with thrombolic risks
* Subjects who weigh less than 40 kg
* Subjects who are pregnant or suspect pregnancy, or subjects who want to become pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Fuji, Principal Investigator — Osaka Kouseinennkin Hospital
Locations (1):
- Osaka, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Fuji T, Fujita S, Kawai Y, Nakamura M, Kimura T, Kiuchi Y, Abe K, Tachibana S. Safety and efficacy of edoxaban in patients undergoing hip fracture surgery. Thromb Res. 2014 Jun;133(6):1016-22. doi: 10.1016/j.thromres.2014.03.009. Epub 2014 Mar 6. PMID 24680549

RESULTS

PARTICIPANT FLOW:
Groups:
- DU-176b: DU-176b oral tablets, 30 mg., taken once daily for 2 weeks
  DU-176b (edoxaban)
- Enoxaparin Sodium: Enoxaparin sodium 20mg(=2000IU)/0.2ml twice daily, subcutaneous injection for 2 weeks
  Enoxaparin sodium 20mg
Period: Overall Study
Arm/Group | DU-176b | Enoxaparin Sodium
Started | 62 | 30
Safety Analysis Population | 59 | 29
Completed | 50 | 26
Not Completed | 12 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Population: Number of baseline participants reflects the safety analysis population
Groups:
- Total: Total of all reporting groups
Arm/Group | DU-176b | Enoxaparin Sodium | Total
Number analyzed (Participants) | 59 | 29 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.5 (11.0) | 75.6 (12.0) | 76.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 22 | 70
  Male | 11 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 59 | 29 | 88
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 59 | 29 | 88

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Major or Clinically Relevant Non-major Bleeding
Description: Bleeding events during the period from the start of treatment with the study drug (study treatment) to the day of the follow-up examination were assessed as the primary endpoints.
Time Frame: 2 weeks
Population: Safety Analysis Set defined as all subjects who were secondarily enrolled in study, but excluded those with significant GCP violations, did not receive any study drug, or had no safety data after start of study treatment. However, subjects who had significant GCP violations, but received at least one dose of study drug, safety data were assessed.
Measure: Number (95% Confidence Interval); unit: percentage of subjects with bleeds
Arm/Group | DU-176b | Enoxaparin Sodium
Number analyzed (Participants) | 59 | 29
percentage of subjects with bleeds | 3.4 [0.9 to 11.4] | 6.9 [1.9 to 22.0]
Statistical Analysis 1: Comparison: DU-176b vs Enoxaparin Sodium; Test type: Superiority or Other; Wilcoxon (Mann-Whitney); Cox Proportional Hazard = -3.5, 95% CI 2-sided [-18.8 to 6.0]

2. Secondary Outcome: Proportion of Subjects With Venous Thromboembolism Events.
Time Frame: 2 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Safety Analysis Set defined as all subjects who were enrolled in the study, but excluded those who had significant GCP violations, who did not receive any doses of the study drug, or who had no safety data after the start of study treatment.
Arm/Group | DU-176b | Enoxaparin Sodium
Serious Adverse Events (participants affected / at risk) | 3/59 | 3/29
Other Adverse Events (participants affected / at risk) | 43/59 | 24/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DU-176b (N=59) | Enoxaparin Sodium (N=29)
postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
fracture displacement (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DU-176b (N=59) | Enoxaparin Sodium (N=29)
cystitis (Infections and infestations) | 3 (3) | 2 (2)
nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2)
urinary tract infection (Infections and infestations) | 7 (7) | 4 (5)
constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
diarrhea (Gastrointestinal disorders) | 3 (4) | 3 (4)
decubitis ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (3)
urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 5 (5)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 3 (3)
blood urine present (Investigations) | 9 (9) | 4 (4)
contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
anal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Blood uric acid increased (Investigations) | 2 (2) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 1 (2)
Eosinophil percentage increased (Investigations) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Investigations) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture displacement (Injury, poisoning and procedural complications) | 2 (2) | 1 (2)
vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Wound haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Chest discomfort (Cardiac disorders) | 2 (2) | 0 (0)
pyrexia (General disorders) | 1 (1) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall not publish the results of the Study at any time without the prior written approval of Sponsor.